CLINICAL TRIAL: NCT05154929
Title: Improving Blood Pressure Control Through the myBPmyLife mHealth Application: A Wearables in Reducing Risk and Enhancing Daily Lifestyle (WIRED-L) Center Study
Brief Title: Improving Blood Pressure Control Through the myBPmyLife mHealth Application
Acronym: myBPmyLife
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Brahmajee K Nallamothu, Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00205845
Record Dates: First submitted 2021-11-30; First posted 2021-12-13 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hypertension
Keywords: high blood pressure; exercise; decrease salty food; smartwatch; mobile application
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Diet; Control Groups

STUDY DESIGN:
Intervention Model Description: This study is a multicenter 6 month randomized controlled clinical trial. This study will investigate the efficacy of two just-in-time adaptive interventions (JITAIs) delivered via a mobile app for patients with hypertension. Eligible participants will be randomized to the two JITAIs or control in a 1:1 manner stratified by site. There will be two sites: the University of Michigan Health System in Ann Arbor and the Hamilton Community Health Network Clinic in Flint.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Other): Participants in the control group will be provided a smartwatch and home blood pressure monitor. They will also be provided with general instructions on how to download and install a physical activity and diet regulation applications (apps) available to the general public. They will still be asked to perform the blood pressure monitoring at regularly scheduled time periods, but do not receive the intervention components notifications in myBPmyLife app developed for the experimental group.
  Interventions: Other: Control Group
- Dietary plus physical activity JITAI (Experimental): Participants in the experimental group will be provided a smarthwatch and home blood pressure monitor. They will then receive the myBPmyLife app that includes push notifications to promote increased physical activity and improve low sodium food choices. The app also provides goal setting for weekly step count and information on low-sodium food choices, as well as feedback on achieving the goals using a dashboard with visualization tools within the mobile application.
  Interventions: Behavioral: Dietary and physical activity JITAI delivered through the myBPmyLife app

INTERVENTIONS:
Behavioral: Dietary and physical activity JITAI delivered through the myBPmyLife app — A Fitbit smartwatch and home blood pressure monitor will be mailed to participants (in both the experimental and control arms). Participants in the intervention arm then will set up and utilize the myBPmyLife app. This app includes push notifications to promote increased physical activity and improve low-sodium food choices, establish goal setting for weekly step count and low sodium food choices, and deliver feedback on achieving the goals using a dashboard visualization within the mobile application.
  Arms: Dietary plus physical activity JITAI
Other: Control Group — Participants will receive the myBPmyLife app, a smartwatch, and blood pressure cuff. The myBPmyLife app will not be fully activated (as they are in the control arm). They will be provided with the option of downloading and installing a mHealth app that is publicly available. In this arm they will also perform the blood pressure monitoring, but do not receive the intervention components through the myBPmyLife app.
  Arms: Control arm

SUMMARY:
This study is enrolling eligible participants that have high blood pressure. Reducing dietary salt intake and engaging in regular physical activity is known to decrease blood pressure in people with hypertension. This trial will determine whether a smartwatch and a mobile health application, which together deliver notifications, can increase activity levels and reduce salt intake for people with high blood pressure. All study activities will be completed online or via a mobile medical application. Participants will not have any face-to-face visits with the study team.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported history of hypertension and no hypertensive medication changes in the last 4 weeks.
* A smartphone with a compatible Apple or Android operating system installed and able to download and use the myBPmyLife app including accepting all permissions
* A valid email address
* Fluent in spoken and written English
* Signed written informed consent. (Note that each participant must be able to consent for themselves.)

Exclusion Criteria:

* Contraindication to performing physical activity or following a sodium restriction diet. The participant must be able to walk and eat on their own without assistive devices.
* Unstable symptoms or markedly elevated BP at enrollment (defined as systolic BP>180 mmHg, diastolic BP>120 millimeters of mercury (mmHg))
* Known secondary causes of hypertension (e.g., adrenal insufficiency, pheochromocytoma), heart failure, or end-stage renal disease
* Difficulty using an upper arm blood pressure cuff due to biceps size or end-stage renal disease or difficulty comfortably wearing a smartwatch
* Wrist too large to wear a smartwatch comfortably.
* Daily sodium intake less than 1500 mg/day as measured by the sodium screener
* Currently pregnant or planning to become pregnant in the next six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2024-01-27 (Actual); Study Completion 2024-01-27 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure between baseline and 6-months | Baseline, 6 months

SECONDARY OUTCOMES:
Number of self-reported low-sodium food choices within 24 hours of a diet notification | within 24 hours of a diet notification
Number of steps taken within 60 minutes of a physical activity notification | within 60 minutes of a physical activity notification
Change in mean daily sodium intake between baseline and 6-months (Block Sodium Screener) | Baseline, up to 6 months
Change in mean daily step count between baseline and 6-months (i.e., 180 days) | Baseline, up to 6 months
Change in diastolic blood pressure from baseline to 6-months (i.e., 180 days) | Baseline, up to 6 months
Trends in weekly systolic BP over the 6-months (i.e., 180 days) | Baseline to weekly assessments that are available up to 24 weeks
Changes in systolic BP from baseline to 60 days, 120 days, and at 180 days (i.e., approximately 2 months) | Baseline, every 60 days from 0 days to 60 days to 120 days to 180 days (i.e., approximately 2 months)
Change in quality-of-life between baseline and 6-months as assessed by the single-item Self-Rated Health (SRH) Questionnaire | Baseline, up to 6 months
  Change in the proportion of SRH responses from baseline to 6-months (i.e., 180 days) across 2 categories: 1) excellent, very good or good versus 2) fair or poor.

CONTACTS AND LOCATIONS:
Overall Officials: Brahmajee K Nallamothu, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Hamilton Community Health Network, Flint, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dorsch MP, Golbus JR, Stevens R, Trumpower B, Basu T, Luff E, Warden K, Giacalone M, Bailey S, Rubick GV, Mishra S, Klasnja P, Newman MW, Skolarus LE, Nallamothu BK. Physical activity and diet just-in-time adaptive intervention to reduce blood pressure: a randomized controlled trial. NPJ Digit Med. 2025 Jul 14;8(1):438. doi: 10.1038/s41746-025-01844-3. PMID 40659778
- [Derived] Golbus JR, Jeganathan VSE, Stevens R, Ekechukwu W, Farhan Z, Contreras R, Rao N, Trumpower B, Basu T, Luff E, Skolarus LE, Newman MW, Nallamothu BK, Dorsch MP. A Physical Activity and Diet Just-in-Time Adaptive Intervention to Reduce Blood Pressure: The myBPmyLife Study Rationale and Design. J Am Heart Assoc. 2024 Jan 16;13(2):e031234. doi: 10.1161/JAHA.123.031234. Epub 2024 Jan 16. PMID 38226507